CLINICAL TRIAL: NCT04316520
Title: A Pilot Study Evaluating the Tolerability of a Ketogenic Diet With Vitamin Supplementation for Patients Receiving Treatment for Metastatic Renal Cell Carcinoma
Brief Title: Ketogenic Diet for Patients Receiving Treatment for Metastatic Renal Cell Carcinoma
Acronym: CETOREIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49RC19_0181
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Renal Cancer
Keywords: metastatic renal cancer; ketogenic diet; immunotherapy; first line treatment; targeted therapy
MeSH Terms: conditions — Kidney Neoplasms | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet (Experimental): Ketogenic diet + standard of care
  Interventions: Dietary Supplement: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Ketogenic diet 2:1
  Other Names: First line treatment

SUMMARY:
The purpose of this study is to evaluate the tolerance of one year of ketogenic diet associated with vitamin supplementation in patients treated for a metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
This research study is a pilot study evaluating the tolerance of a ketogenic diet associated with a standard of care in patient with metastatic renal cell carcinoma.

The drugs involved in this study could be NIVOLUMAB + IPILIMUMAB, PEMBROLIZUMAB + AXITINIB, SUNITINIB or PAZOPANIB.

Cancer cells are known to have an increased glycolytic activity that allows them to product energy from anaerobic degradation of glucose. A ketogenic diet places the body in ketosis state. It forces the body to burn fat instead of glucose. Fat metabolism occurs via the mitochondrial oxidative phosphorylation. By reducing sugar intake and regulating energy metabolism, the ketogenic diet could contribute to limit tumor progression.

This diet will be introduced during one year, patient will be monitored closely with biological tests and radiological assessments every three month.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with histologically-confirmed renal cell carcinoma
2. At least one CT-verified metastasis ≥ 10 mm, not previously irradiated
3. Treatment : PAZOPANIB, SUNITINIB, PEMBROLIZUMAB/AXITINIB or NIVOLUMAB/IPILIMUMAB (for first line), NIVOLUMAB, CABOZANTINIB, AXITINIB, SORAFENIB, TKI anti-VEGF, other therapy for second and third line of treatment
4. Men and women, aged ≥ 18 years
5. OMS ≤ 1
6. Screening laboratory values must meet the following criteria and should be obtained prior to commencement of treatment:

   1. Hemoglobin ≥ 9 g/dL, neutrophils ≥ 1000 /mm3, platelets ≥ 100 000 /mm3, leukocytes ≥ 2000 /mm3
   2. Total bilirubin ≤ 1,5 ULN, ASAT and ALAT ≤ 3 x ULN
   3. Creatinine clearance ≥ 30 mL/min, verified proteinuria above or equal to 1g/24 hours measured from 24 hours of urine if the urinary protein
   4. Corrected calcium ≤ ULN
7. Patient must have signed and dated informed consent
8. Patient must have an internet connection

Exclusion Criteria:

1. Any contraindication to a ketogenic diet : primary carnitine deficiency, fatty acid beta-oxidation and cytogenesis deficiencies, pyruvate carboxylate deficiency, porphyria
2. Swallowing disorder
3. Important surgical procedure within the 4 weeks before treatment
4. Prior radiotherapy must have been completed at least 2 weeks prior to treatment
5. Pregnant women or breastfeeding
6. Subjects with previous malignancies (except non-melanoma skin cancer and the following endometrial in situ cancers) are excluded unless a complete remission was achieved at least 3 years prior to study entry and no additional therapy is required during the study period
7. Subjects with symptomatics brain metastases, uncontrolled compression of the spinal cord, carcinomatous meningitis, signs of cerebral or leptomeningeal involvement
8. Uncontrolled blood pressure (SBP >150 mmH et DBP >100 mmHg)
9. Any serious or uncontrolled medical disorder during the last 6 months : hepatic insufficiency, renal insufficiency, respiratory insufficiency
10. Patients with any severe medical conditions within 6 month prior to inclusion such as : myocardial infarction, severe/instable angina pectoris, coronary artery bypass surgery, NYHA III or IV congestive heart failure, stroke or transient ischemic attack
11. Patients with sere medical conditions within 3 month prior to inclusion such as : grade 3 or grade 4 gastrointestinal bleeding, peptic ulcer treatment resistant, esophagitis or ulcerated gastritis, infectious or inflammatory bowel disease, diverticulitis, thrombosis, pulmonary embolism or other uncontrolled thromboembolic event, unhealed bone fractures
12. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
13. Malabsorption syndrome
14. Uncontrolled infection
15. QT/QTc interval > 450 msec for men and > 470 msec for women
16. Concomitant treatments : strong inducers of CYP3A4 (DEXAMETHASONE, PHENYTOINE, CARBAMAZEPINE, RIFAMPICINE, RIFABUTINE, RIFAPENTINE, PHENOBARBITAL, and ST. JOHN'S WORT)
17. Social, psychological or medical condition that may interfere with participation in the study or its evaluation
18. Patient deprived of liberty by judicial or administrative decision
19. Patient with psychiatric treatment under duress
20. Patient subject to legal protection measures
21. Patient unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Tolerance of one year of ketogenic diet 2:1 | 1 year
  Frequency of adverse events evaluation

SECONDARY OUTCOMES:
Compliance of ketogenic diet | 1 year
  Pourcentage of compliant patients
Progression free survival according to RECIST 1.1 at 2 years | 2 years
  Assessed by RECIST 1.1
Overall survival at 2 years | 2 years
  Assessed by RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No